CLINICAL TRIAL: NCT04014569
Title: Determination of Automated Multiple Insulin Dose Injections Settings Using the MDI/SMBG Advisor for Patients With Type 1 Diabetes -Data Collection, Observational & Proof of Concept Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators decision
Sponsor: Rabin Medical Center (Other)
Collaborators: DreaMed (Industry); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC018718ctil
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes; Multiple Daily Injections
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MPSA Algorithm (Experimental): Insulin dosing will be adjusted using the MPSA algorithm
  Interventions: Device: MPSA Algorithm

INTERVENTIONS:
Device: MPSA Algorithm — Insulin dosing will be adjusted using the MPSA Algorithm

SUMMARY:
The MDI (Multiple Daily Injections) plus SMBG |(Self Monitoring Blood Glucose) Advisor (MPSA) is a software product that is designed to assist in insulin dosage decision making for subjects with T1DM using multiple daily injection and SMBG.

The study will focus on the development, validation and eventually testing of the MPSA algorithm use. The major objective of the project is to develop an algorithm that will be able to optimize treatment plan parameters of MDI patients who use SMBG as glucose monitoring method. The clinical study has two segments. Segment A is an observational study needed for the development of the algorithm (this segment was already completed at the time of the registration) and Segment B is a proof of concept interventional study to validate the algorithm's Safety and Efficacy.

Up to 20 patients using MDI and SMBG or Flash Glucose Monitoring (FGM) without using glucose trends will be enrolled to this proof of concept study. The study will evaluate the algorithm use for a period of 11 weeks. Post screening, patients will undergo a two weeks run-in period while using MDI and SMBG or FGM (patients that do not use FGM will be provided with blinded Libre Flash to be used during the run-in period and 2 weeks prior to arriving to end of study visit). Then, patients will undergo insulin treatment plan changes every week for 7 weeks. At the first 3 weeks insulin dose adjustments will be done for basal insulin dose only, week 4 will be without changes, and in the next 3 weeks the carbohydrate ratio will be amended. No recommendations will be given during the last two weeks of the study. These two weeks will be used for data analysis. Each recommendation of the Advisor will be approved by a physician before implementation. Glucose outcomes will be evaluated comparing the two weeks run-in period to the last two weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented T1D for at least 1 year prior to study enrolment
* Subjects aged ≥ 14 years and up to 30 years
* A1c at inclusion ≥ 7 % and ≤ 10%
* Using MDI of Basal/bolus therapy - basal insulin either Glargine/Lantus or Tregludec insulin and bolus short acting insulin analogs either aspart/Novorapid or Lispro/Humalog
* Using SMBG or flash glucose monitoring (FGM/Libre) without using glucose trends
* BMI SDS - below the 97th percentile for age
* Subjects willing to follow study instructions

Exclusion Criteria:

* An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment
* Concomitant diseases/ treatment that influence metabolic control or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety
* Participation in any other interventional study
* Known or suspected allergy to trial products
* Female subject who is pregnant or planning to become pregnant within the planned study duration
* Subject needs to travel by air during the study duration

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of sensor glucose readings within range of 70-180 mg/dl | Final visit (day 42)

SECONDARY OUTCOMES:
Percentage of sensor glucose readings below 54 mg/dl | Final visit (day 42)
HbA1c | Final visit (day 42)
Number of Severe Hypoglycemia events | Final visit (day 42)
Number of Diabetic Ketoacidosis events | Final visit (day 42)

OTHER OUTCOMES:
Percentage of sensor glucose readings below 70 mg/dl | Final visit (day 42)
Percentage of sensor glucose readings below 50mg/dl | Final visit (day 42)
Percentage of sensor glucose readings above 180mg/dl | Final visit (day 42)
Percentage of sensor glucose readings above 250mg/dl | Final visit (day 42)
Number of unexplained hyperglycemic events | Final visit (day42)
Area above the curve of 180mg/dl | Final visit (day 42)
Area above the curve >180mg/dl | Final visit (day 42)
Area under the curve of 70mg/dl | Final visit (day 42)
Area under the curve <70mg/dl | Final visit (day 42)
Mean sensor blood glucose | Final visit (day42)
Glucose variability measured by SD (standard deviation) | Final visit (day 42)
Number of recommendations for changes in settings per patient | Final visit (day 42)
Number of recommendations for changes in setting per iteration | Final visit (day 42)
Number of physician override advisor recommendations | Final visit (day 42)

CONTACTS AND LOCATIONS:
Locations (1):
- Schnider children medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No